CLINICAL TRIAL: NCT06827301
Title: Transcutaneous Auricular Vagus Nerve Stimulation Combined With Rehabilitation Therapy for the Treatment of Post-stroke Dysphagia
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation for Treating Post-stroke Dysphagia
Acronym: LOGIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Di Lazzaro Vincenzo, Prof, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOGIC
Record Dates: First submitted 2024-12-02; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Dysphagia Following Cerebrovascular Accident
Keywords: vagus nerve stimulation; dysphagia; stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real t-VNS (Experimental): real t-VNS on left ear for 40 minutes, daily for 3 consecutive days, simultaneously with speech therapy.
  Interventions: Device: Non Invasive vagus nerve stimulation
- Sham t-VNS (Active Comparator): sham t-VNS on left ear for 40 minutes, daily for 3 consecutive days, simultaneously with speech therapy.
  Interventions: Device: Non Invasive vagus nerve stimulation

INTERVENTIONS:
Device: Non Invasive vagus nerve stimulation — Transcutaneous Auricular Vagus Nerve Stimulation

SUMMARY:
The aim of the present project is to use transcutaneous auricular vagus nerve stimulation (t-VNS) for the treatment of dysphagia in acute stroke patients to improve swallowing function and reduce mortality and disability related to this condition.

30 patients will be randomized into one of the two arms of the study:

* REAL: real t-VNS + speech therapy
* SHAM: t-VNS placebo + speech therapy. The experimental treatment consists in the association between t-VNS (real or placebo) and speech therapy exercises to improve swallowing functionality. Each patient will undergo a speech therapy rehabilitation session lasting approximately 40 minutes a day for 3 consecutive days, simultaneously with t-VNS on left ear.

Swallowing function and clinical conditions will be evaluated before the intervention (baseline, T0), immediately after the intervention (T1) and 3 months after the intervention (T2).

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic or hemorrhagic stroke (within 7 days of onset)
* Dysphagia diagnosed by FEES with a Fiberoptic Endoscopic Dysphagia Severity Scale (FEDSS) score between 3 and 5

Exclusion criteria:

* Pre-existing stroke dysphagia
* Dementia or other medical conditions that may interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Swallowing function | Baseline, Immediately after intervention
  Swallowing video fluoroscopic will be used to measure swallowing function

SECONDARY OUTCOMES:
Disability | Baseline, Immediately after intervention, 3 months after intervention
  Disability will be measured by mRS and the necessity of nasogastric tube/gastrostomy.
Mortality | Baseline, Immediately after intervention, 3 months after intervention
  Number of deaths
Morbidity | Baseline, Immediately after intervention, 3 months after intervention
  Number of aspiration pneumonia
Swallowing function | Baseline, 3 months after intervention
  Swallowing video fluoroscopic will be used to measure swallowing function

CONTACTS AND LOCATIONS:
Locations (1):
- Università Campus Bio-Medico di Roma, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided